CLINICAL TRIAL: NCT03606161
Title: Feasibility of Navigated Repetitive Transcranial Magnetic Stimulation (nrTMS) to Augment the Effects of Motor Rehabilitation in Brain Tumor Patients
Brief Title: Navigated Repetitive Transcranial Magnetic Stimulation in Improving Motor Rehabilitation in Participants With Brain Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0269; NCI-2018-01476 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0269 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (nrTMS) (Experimental): Between 1-7 days after standard of care surgery, participants undergo 10 nrTMS sessions over 30 minutes each over 3 weeks.
  Interventions: Other: Questionnaire Administration; Procedure: Transcranial Magnetic Stimulation

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Procedure: Transcranial Magnetic Stimulation — Undergo nrTMS
  Other Names: TMS

SUMMARY:
This trial studies how well navigated repetitive transcranial magnetic stimulation works in improving motor rehabilitation in participants with brain tumors. Navigated repetitive transcranial magnetic stimulation may help improve patients' lost motor function after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine feasibility of conducting 10 sessions of navigated repetitive transcranial magnetic stimulation (nrTMS) during the post-surgical rehabilitation time period.

EXPLORATORY OBJECTIVES:

I. Explore the effects of the nrTMS training program on motor recovery. II. Explore changes in cortical activity: electroencephalographic (EEG) activity including event-related potentials (ERPs) and motor evoked potentials (MEPs) will be assessed from baseline to end of treatment (EOT).

OUTLINE:

Between 1-7 days after standard of care surgery, participants undergo 10 nrTMS sessions over 30 minutes each over 3 weeks.

After completion of study, participants are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain tumors associated with the motor cortex
* Understand and read English, sign a written informed consent, and be willing to follow protocol requirements
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Motor impairment must be related to the surgical procedure or the tumor itself (in the opinion of the treating physician)
* Patients who are within 7 days of brain tumor resection associated with the motor cortex
* Eligibility for the nrTMS treatment will be based on motor ability and will be determined postoperatively by the surgeon

Exclusion Criteria:

* Patients who are taking any antipsychotic medications
* Patients who have ever been diagnosed with bipolar disorder or schizophrenia
* Patients with a history of stroke

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention adherence | Up to 3 months
  Will be defined as a participant as completing at least 70% of the (i.e., seven out of 10) treatment sessions. Feasibility will be defined as: 1) at least 70% of the participants adhere to the treatment. Patients will have to finish all 10 trains in each navigated repetitive transcranial magnetic stimulation (nrTMS) run in order to be considered complete; 2) at least 37% of the eligible patients (at a rate of approximately 3/8 per month) enroll in the study.

OTHER OUTCOMES:
Motor recovery | Up to 3 months
  Will conduct a paired sample t-test, subtracting post-intervention scores from pre-intervention scores at each post-intervention time point.
Changes in cortical activity | Baseline up to 3 months
  Will include pre and post comparisons of the electroencephalogram, via event related potential (ERP) analysis. Baseline LORETA analyses will include global differences in cortical activation as well as site-specific dominant frequencies for each patient. Will observe baseline differences in amplitude, power, and relative power for delta, theta, alpha, low beta, high beta, gamma, theta/beta ratio, and alpha/beta ratios for each patient. ERP analysis will compare amplitudes in the surgical hemisphere and the normal hemisphere via an asymmetry index which will be computed for each pair of homologous electrodes and in each condition: AI = (surgical ERP) - (healthy ERP on the homologous site)/the peak ERP at any site. To assess inter-hemispheric imbalances in cortical excitability, will determine differences in the nrTMS group and the Human Brain Index Reference Database (HBIRD).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Prinsloo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org